CLINICAL TRIAL: NCT04359459
Title: Nasal CIliated EPithelial Genetic And Single Cell RNA prOfiLes of miLd, Severe and Very Severe COVID-Nineteen patIents (CIPOLLINI) Study
Brief Title: Nasal Epithelial Genetic and Single Cell RNA COVID-19 Study
Acronym: CIPOLLINI
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19 pandemie ended
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, MD PhD, University Medical Center Groningen
Other Study IDs: CIPOLLINI
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood sampling: 1x serum, 1x plasma + buffycoat, 1x protease inhibitor tube, 1x PAXgene RNA tube
  * Nasal brushes: 5 nasal brushes will be collected, 1x RNAProtect Cell solution, 2x 10Xgenomic (single cell sequencing), 1 x DNA methylation in empty tube, 1 x in 2mL universal virus transport medium.
  * Stool sample - 1 tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild COVID-19: Patients with mild disease who tested positively for SARS-CoV2 infection, but only experience mild symptoms and do not need hospitalization.
- Severe COVID-19: Patients with severe disease admitted to hospital, without the need to be admitted to the intensive care.
- Very Severe COVID-19: Patients with very severe disease admitted to intensive care, who require mechanical ventilation.

SUMMARY:
Rationale:

The investigators hypothesize that genetics and the nasal epithelial response to SARS-CoV2 are critical determinants of the immune response to viral infection, and predict clinical outcome in COVID-19 patients.

Objective:

The main objective is to assess whether genetic background and/or the nasal epithelial gene expression in response to SARS-CoV2 is different in patients with mild, severe or very severe disease. The secondary goal of this study is to investigate a) the role of the ACE2-AngII system during SARS-CoV2 in relation to outcome b) the long-term consequences of mild, severe, and very severe COVID-19 infection c) the association between mild, severe and very severe COVID-19 with clinical & molecular markers of disease progression d) whether the faeces microbiome, virome or metabolomics profile predicts clinical outcome in COVID-19 patients and e) to investigate whether pre-existing antibodies towards other coronaviruses play a role in severe disease development.

Study design:

Prospective open label clinical observational study. In this study samples will be collected from 150 COVI-19 patients ( 50 mild (group 1), 50 severe (group 2) and 50 very severe (group 3) ). Blood, nasal brushes and stool will be collected for all groups at hospital admission and 3 months after recovery, and for groups 2 & 3 at day 3, at day 14, and before detubation

Study population:

A total of 150 patients diagnosed with COVID-19 will be included. The investigators aim for 50 patients per group, divided over 3 groups:

Group 1 Patients with mild disease who tested positively for SARS-CoV2 infection, but only experience mild symptoms and do not need hospitalization.

Group 2 Patients with severe disease admitted to hospital, without the need to be admitted to the intensive care.

Group 3 Patients with very severe disease admitted to intensive care, who require mechanical ventilation.

Main study parameters/endpoints:

The primary endpoint of this study is the identification of genes, pathways and cell populations that associate with clinical outcome and disease progression in mild, severe and very severe COVID-19 patients.

DETAILED DESCRIPTION:
Rationale:

The currently ongoing world-crippling pandemic with the new SARS-CoV2 virus shows the desperate and urgent need for a better understanding of the biological pathways activated by the virus inducing Coronavirus disease 2019 (COVID-19) in infected patients. A subset of COVID-19 patients develop very severe respiratory symptoms requiring hospital admission with or without the need for mechanical ventilation, whereas others experience mild flu-like symptoms. The biological mechanisms underlying this striking difference in clinical outcome and the long term consequences are unknown, yet a genetic factor seems likely. SARS-CoV2 enters cells via the ACE2 receptor and the activating protease TMPRSS2 which have recently been shown to be strongly enriched in nasal epithelium. The investigators hypothesize that genetics and the nasal epithelial response to SARS-CoV2 are critical determinants of the immune response to viral infection, and predict clinical outcome in COVID-19 patients.

Objective:

The main objective is to assess whether genetic background and/or the nasal epithelial gene expression in response to SARS-CoV2 is different in patients with mild, severe or very severe disease. The secondary goal of this study is to investigate a) the role of the ACE2-AngII system during SARS-CoV2 in relation to outcome b) the long-term consequences of mild, severe, and very severe COVID-19 infection c) the association between mild, severe and very severe COVID-19 with clinical & molecular markers of disease progression d) whether the faeces microbiome, virome or metabolomics profile predicts clinical outcome in COVID-19 patients and e) to investigate whether pre-existing antibodies towards other coronaviruses play a role in severe disease development.

Study design:

Prospective open label clinical observational study. In this study samples will be collected from 150 COVI-19 patients ( 50 mild (group 1), 50 severe (group 2) and 50 very severe (group 3) ). Blood, nasal brushes and stool will be collected for all groups at hospital admission and 3 months after recovery, and for groups 2 & 3 at day 3, at day 14, and before detubation. Study subjects will be retrospectively allocated to the groups.

Study population:

A total of 150 patients diagnosed with COVID-19 will be included. The investigators aim for 50 patients per group, divided over 3 groups:

Group 1 Patients with mild disease who tested positively for SARS-CoV2 infection, but only experience mild symptoms and do not need hospitalization.

Group 2 Patients with severe disease admitted to hospital, without the need to be admitted to the intensive care.

Group 3 Patients with very severe disease admitted to intensive care, who require mechanical ventilation.

Main study parameters/endpoints:

The primary endpoint of this study is the identification of genes, pathways and cell populations that associate with clinical outcome and disease progression in mild, severe and very severe COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have to be tested (PCR) positive for SARS-CoV2 infection.
2. Provided written informed consent

Exclusion Criteria:

1. No comprehension of Dutch or English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1 Patients with mild disease who tested positively for SARS-CoV2 infection, but only experience mild symptoms and do not need hospitalization.
  Group 2 Patients with severe disease admitted to hospital, without the need to be admitted to the intensive care.
  Group 3 Patients with very severe disease admitted to intensive care, who require mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Nasal epithelial transcriptional response to SARS-CoV2 | Observational-baseline
  To assess how the nasal epithelial transcriptional response to SARS-CoV2 is different in patients with mild, severe, or very severe disease.

SECONDARY OUTCOMES:
ACE2-AngII system | Observational-baseline
  To assess the role of the ACE2-AngII system during SARS-CoV2 in relation to disease outcome (mild, severe, very severy COVID)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — UMCG, Department of pulmonology; Janesh Pillay, MD PhD, Principal Investigator — UMCG, Intensive Care Medicine

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on request.